CLINICAL TRIAL: NCT01670396
Title: G Protein β3 Subunit (GNB3) Polymorphism and Restenosis of Coronary Drug-eluting Stents
Brief Title: Genetics Study of In-stent Restenosis
Acronym: ISR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZS-XN-ISR
Record Dates: First submitted 2012-08-15; First posted 2012-08-22 (Estimated); Last update posted 2012-08-22 (Estimated); Status verified 2012-08

CONDITIONS: Coronary Artery Disease
Keywords: coronary stent implant; polymorphism; G protein; drug-eluting stent; restenosis
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- in-stent restenosis
- non-in-stent restenosis

SUMMARY:
The investigators hypothesized that genetic variants of G protein influence the development of restenosis and clinical outcome of patients receiving drug-eluting stents (DES).

DETAILED DESCRIPTION:
Although drug-eluting stents (DES) have reduced restenosis rates compared with bare-metal stents, the restenosis rate is still high in the high-risk group. G protein plays important roles in the signal transduction leading to vascular smooth muscle proliferation. The initial and subsequent studies suggest that the T allele of C825T polymorphism is associated with enhanced transmembrane signaling via Gi proteins.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent follow-up angiography. All the patients must had been implanted with DES during the last two years.

Exclusion Criteria:

* For the non-ISR group, the patients underwent follow-up angiography less than 6 months away from stent implanting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2012-03; Primary Completion 2012-08 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
In-stent restenosis | 6-24months after stent implanting

SECONDARY OUTCOMES:
target lesion revascularization (TLR) | 6-24months after stent implanting
re-myocardial infarction | 6-24months after stent implating

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Shanghai, China